CLINICAL TRIAL: NCT00879541
Title: A Phase II, Multicentre, Double-blinded, Randomised, Cross-over Study to Evaluate Efficacy, Safety and Pharmacokinetics of Biostate® in Subjects With Haemophilia A.
Brief Title: Study of a pd vWF/FVIII, Biostate®, in Subjects With Haemophilia A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Global Head Clinical Research & Development, CSL Behring
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CSLCT-BIO-07-47; 1472 (Other: CSL Behring)
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; von Willebrand Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PK Biostate® [SP] (Other): Part 1: PK subjects are randomized to receive Biostate® [SP] either on Day 1 or Day 8.
  Part 3: All PK subjects receive Biostate® [SP] on Day 180.
  Interventions: Biological: Biostate® [SP]
- PK Biostate® [RP] (Other): Part 1: PK subjects are randomized to receive Biostate® [RP] either on Day 1 or Day 8.
  Interventions: Biological: Biostate® [RP]
- Efficacy (Experimental): Part 2: This arm includes all subjects during the efficacy component of the study.
  Interventions: Biological: Biostate® [SP]

INTERVENTIONS:
Biological: Biostate® [SP] — Single bolus intravenous dose of 50 IU/kg
  Other Names: Human Coagulation Factor VIII / von Willebrand Factor
  Arms: PK Biostate® [SP]
Biological: Biostate® [SP] — The dose is dependent on the reason for use and may consist of repeated bolus doses as required to manage haemophilia condition.
  Other Names: Human Coagulation Factor VIII / von Willebrand Factor
  Arms: Efficacy
Biological: Biostate® [RP] — Single bolus intravenous dose of 50 IU/kg.
  Other Names: Biostate®; Human Coagulation Factor VIII / von Willebrand Factor
  Arms: PK Biostate® [RP]

SUMMARY:
The aim of this study are to

* assess the efficacy of Biostate® [Study Product (SP)] in subjects with Haemophilia A
* compare the pharmacokinetics of Biostate® [SP] with the previously marketed product Biostate® (here referred to as Biostate® [Reference Product (RP)]).

This study is divided into 3 parts:

Part 1: Cross-over pharmacokinetic (PK) component. PK subjects will be randomised to determine the order in which they receive the two study products. This part of the study is double-blinded.

Part 2: Efficacy component. All subjects will receive Biostate® [SP] as required to manage their haemophilia condition for an estimated period of 6 months (or minimum of 50 exposure days) to assess efficacy and safety of the product. This part of the study is open-label.

Part 3: Repeat pharmacokinetic assessment. Subjects who participated in Part 1 (PK component) will undergo a repeat PK assessment on Day 180 following administration of Biostate® [SP].

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Haemophilia A with ≤ 1% Factor VIII (FVIII) levels in the absence of factor replacement
* Evidence of vaccination against hepatitis A and B (or presence of antibodies against hepatitis A and B due to either a previous infection or prior immunisation) within 10 years prior to Day 1 documented in the medical notes
* At least 150 days of prior exposure to a FVIII replacement product
* Written informed consent given

Exclusion Criteria (for participation in the pharmacokinetic (PK) component):

* Active bleeding
* Body weight > 100 kg

Exclusion Criteria (for all subjects):

* Receipt of an infusion of any FVIII product, cryoprecipitate, whole blood, plasma, or desmopressin acetate (DDAVP) in the 4 days prior to Day 1
* Known history of FVIII inhibitors, or FVIII inhibitor level > 0.6 Bethesda Units (BU) at screening
* Receipt of aspirin or other Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) within 7 days of administration of study product.
* CD4 lymphocytes < 200/µL. Subjects wo are HIV-1 positive may be considered for the study if viral load ≤ 200 particles/µL at screening and all other eligibility criteria are met.
* Impaired liver function ie. bilirubin >1.5 x upper limit of normal (ULN) and/or AST/ALT > 2.5 x ULN at screening.
* Acute or chronic medical condition, other than haemophilia A, which may, in the opinion of the Investigator, affect the conduct of the study
* von Willebrand Disease (VWD) with Von Willebrand Factor:Ristocetin Cofactor (vWF:RCo) level < 50 IU/dL at screening
* Evidence or a history (within the previous 12 months) of abuse of any drug substance, licit or illicit
* Known or suspected hypersensitivity or previous evidence of severe side effects to Biostate®, FVIII concentrates or human albumin
* Participation in a clinical study or use of an investigational compound (e.g. a new chemical entity not approved for clinical use) in the 3 months preceding the first day of study drug administration, or plans to enter such a study during the study period
* Not willing and/or not able to comply with study requirements

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Haemostatic efficacy | Monthly, until final study visit
Number of treatments/units required to resolve any bleeding event | From Day 1 until final study visit
FVIII concentrate usage (number of infusions, IU/kg per event, per month, and per year) | From Day 1 until final study visit
Assessment of blood loss during any surgical procedure | From Day 1 until final study visit
Pharmacokinetics of FVIII activity | Up to 48 hours following infusions (Part 1 and Part 3 only)

SECONDARY OUTCOMES:
The nature, frequency and incidence of adverse events | From Day 1 until final study visit
Development of FVIII inhibitors | From Day 1 until final study visit

CONTACTS AND LOCATIONS:
Locations (14):
- Bulgaria (3):
  - Study Site, Plovdiv
  - Study Site, Sofia
  - Study Site, Varna
- Study Site, Skopje, North Macedonia
- Poland (7):
  - Study Site, Bialystok
  - Study Site, Gdansk
  - Study Site, Krakow
  - Study Site, Lublin
  - Study Site, Poznan
  - Study Site, Warsaw
  - Study Site, Wroclaw
- Russia (3):
  - Study Site, Barnaul
  - Study Site, Kirov
  - Study Site, Moscow